CLINICAL TRIAL: NCT06006923
Title: Randomized Trial of Regorafenib in Combination With Pembrolizumab or Pembrolizumab Monotherapy With an Efficacy Lead-in of Regorafenib and Pembrolizumab for Patients With MSI-H Colorectal Cancer
Brief Title: Regorafenib in Combination With Pembrolizumab or Pembrolizumab for MSI-H Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated per directive from Bayer due to funding.
Sponsor: Anwaar Saeed (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Anwaar Saeed, Associate Professor of Medicine, Chief, Gastrointestinal Medical Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCC 23-041
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: MSI-H Colorectal Cancer
Keywords: multi-kinase inhibitor; receptor tyrosine kinases; anti-PD1 blockade; immune checkpoint inhibitor; vascular endothelial growth factor receptor (VEGFR)
MeSH Terms: interventions — regorafenib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pembrolizumab + Regorafenib (Experimental): Pembrolizumab: 200mg, Q3 weeks
  Regorafenib: 60mg Cycle 1 Day 1 90 mg Cycle 2 Day 1
  Interventions: Drug: Regorafenib; Drug: Pembrolizumab
- Pembrolizumab (Active Comparator): Pembrolizumab: 200mg, Q3 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Regorafenib — A multi-kinase inhibitor that targets several receptor tyrosine kinases including vascular endothelial growth factor receptor (VEGFR), which may also have immunomodulatory affect in the tumor microenvironment.
  Other Names: BAY 73-4506; Stivarga
  Arms: Pembrolizumab + Regorafenib
Drug: Pembrolizumab — An anti-PD1 blockade / immune checkpoint inhibitor treatment approved for patients with high microsatellite instability (MSI-H) colorectal cancer (CRC) as first line therapy.
  Other Names: Keytruda

SUMMARY:
This is a trial of Regorafenib in combination with pembrolizumab for patients with MSI-H colorectal cancer consisting of lead-in phase examining preliminary efficacy and safety, followed by a randomized phase to further examine efficacy.

DETAILED DESCRIPTION:
Regorafenib is a multi-kinase inhibitor that targets several receptor tyrosine kinases including vascular endothelial growth factor receptor (VEGFR). Regorafenib may also have immunomodulatory affect in the tumor microenvironment. Preclinical and early clinical studies indicate there is a potential for synergistic activity of regorafenib with immune checkpoint inhibitors that can be leveraged to augment antitumor immunity. Pembrolizumab, anti-PD1 blockade, has been approved for patients with high microsatellite instability (MSI-H) colorectal cancer (CRC) as first line therapy. However, there is still an unmet need to enhance the efficacy of immune checkpoint inhibitors for patients with MSI-H colorectal cancer. The efficacy of TKI and immune checkpoint inhibitor combination have been shown in clinical studies for solid tumors particularly for those that are responsive to immune checkpoint inhibitors therapy. Therefore, there is strong rationale for the combination of regorafenib and pembrolizumab in MSI-H colorectal cancer in which there is increased VEGF activity compared to MSS counterpart. A recent retrospective study showed significantly improved response to regorafenib among patients with MSI-H colorectal cancer, compared to patients with MSS colorectal cancer. Collectively, this combination may increase anti-tumor immune response and clinical effectiveness of immunotherapy for patients with MSI-H colorectal cancer. Based on prior clinical trials, the target regorafenib dose in this study is determined to be 90 mg. However, patients in the lead-in phase will receive regorafenib 60 mg in combination with 200mg of pembrolizumab Q3 weeks in the first cycle to increase tolerance and study compliance. The dose of regorafenib will be increased to 90 mg by Cycle 2. An interim analysis will be performed after completion of data collection for the lead-in phase. Target enrollment for the lead-in phase is approximately 22 patients. Following the futility analysis in lead-in phase, the randomized phase target enrollment is determined to be 66 patients per arm, for a total trial enrollment of 154 participants. Patients who received 3 or less cycles of chemotherapy prior to the determination of MMR-D and MSI-H disease can be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed mismatch repair deficient or microsatellite instability high advanced stage colorectal cancer
2. Measurable disease (per RECIST v1.1)
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
4. Age > 18
5. The patient must be able to swallow oral medication.
6. Adequate organ function based on the following lab assessments:

   1. ANC must be ≥ 1500/mm3
   2. platelet count must be ≥ 100,000/mm3
   3. WBC count ≥ 2.5 × 109 /L
   4. Hemoglobin must be ≥ 9 g/dL
   5. Alkaline phosphatase ≤ 2.5× upper limit of normal (ULN) with the exception of patients with documented liver or bone metastases who should have ALP ≤ 5.0× ULN
   6. AST and ALT ≤ 2.5× ULN with the exception of patients with documented liver metastases who may have AST and/or ALT ≤ 5.0× ULN
   7. International normalized ratio (INR) ≤ 1.5 x ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless receiving treatment with therapeutic anticoagulation
   8. Total bilirubin ≤ 1.5× ULN (≤ 3× ULN if Gilbert syndrome present)
   9. Serum albumin ≥ 2.8 g/dL or 28 g/L
   10. Creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula) or creatinine ≤ 1.5× ULN
7. No more than three cycles of prior fluoropyrimidine-based chemotherapy including folinic acid, fluorouracil, and oxaliplatin (FOLFOX); folinic acid, fluorouracil, and irinotecan (FOLFIRI); and, folinic acid, fluorouracil, oxaliplatin, and irinotecan (FOLFOXIRI) excluding adjuvant treatment
8. Patients (male or female) of reproductive potential must agree to use an effective method of contraception (as discussed with treating physician) from the time consent is signed, during study therapy, and for at least 8 weeks after the last dose of study therapy.
9. Patients who received no more than 1 cycle of pembrolizumab monotherapy will be still eligible to be enrolled in lead in phase of the trial

Exclusion Criteria:

1. Prior anti-programmed death 1 (anti-PD-1) or anti-cytotoxic T-lymphocyte-associated antigen 4 (anti-CTLA-4) based therapy
2. More than 3 cycles of chemotherapy or progression of disease on first line therapy excluding adjuvant treatment and any systemic anticancer treatment within 2 weeks or 5 half-lives (whichever is shorter) prior to start of study treatment
3. Active autoimmune disease
4. Pregnant or lactating females
5. Uncontrolled human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV); patients with undetectable viral load and CD4 count > 200 will be eligible for enrollment
6. Active untreated brain metastasis
7. Uncontrolled hypertension (HTN: systolic pressure > 150 mmHg or diastolic pressure > 90 mmHg on repeated measurements) and cardiovascular events within 12 months of start of treatment
8. Active infection or chronic infection requiring chronic suppressive antibiotics
9. No active cancer such as colon cancer other than adenocarcinoma (e.g., sarcoma, lymphoma, carcinoid) within 1 year
10. Patients with severe hepatic impairment (Child-Pugh C) are excluded as regorafenib has not been studied in this population and exposure might be increased in these patients
11. Major surgical procedure or significant traumatic injury within 28 days before start of study medication
12. Non-healing wound, non-healing ulcer, or non-healing bone fracture
13. Patients with evidence or history of any bleeding diathesis, irrespective of severity
14. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication:

    1. Major surgical procedure or significant traumatic injury within 28 days before start of study medication
    2. Non-healing wound, non-healing ulcer, or non-healing bone fracture
    3. Patients with evidence or history of any bleeding diathesis, irrespective of severity
    4. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR), Lead-in Phase | Up to 12 months (lead-in phase)
  Percentage of patients with partial response (PR) or complete response (CR) to the treatment per RECIST 1.1. criteria. v1.1. Per RECIST v1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or nontarget) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free Survival (PFS), Randomize Phase | Up to 24 months
  Median number of months from time of randomization to the date of disease progression or death from any cause. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events Related to Treatment | Up to 24 months (lead-in phase)
  Percentage of patients that experience Adverse Events (AEs) and/or Serious Adverse Events (SAEs) related to study treatment, per NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0. The maximum grade for each type of toxicity will be recorded for each patient.
Adverse Events and Serious Adverse Events Related to Treatment | Up to 24 months (beginning at start of post lead-in phase)
  Percentage of patients that experience Adverse Events (AEs) and/or Serious Adverse Events (SAEs) related to study treatment, per NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0. The maximum grade for each type of toxicity will be recorded for each patient.
Progression-free Survival (PFS), Lead-In Phase | Up to 24 months
  Median number of months from time of randomization to the date of disease progression or death from any cause. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Overall Survival (OS) | Up to 48 months (lead-in phase)
  Median number of months from start of treatment to death from any cause.
Overall Survival (OS) | Up to 24 months (beginning at start of post lead-in phase)
  Median number of months from time of randomization to death from any cause.
Objective Response Rate (ORR), Randomized Phase | Up to 12 months (beginning at start of post lead-in phase)
  Percentage of patients with partial response (PR) or complete response (CR) to the treatment per RECIST 1.1. criteria. v1.1. Per RECIST v1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or nontarget) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Anwaar H Saeed, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No